CLINICAL TRIAL: NCT03903900
Title: Redesign of Everyday Activities and Lifestyle With Occupational Therapy for Chronic Pain Patients - A Feasibility Study of an Occupational Therapy Intervention Added a Multidisciplinary Biopsychosocial Treatment at a Danish Pain Centre
Brief Title: Redesign of Everyday Activities and Lifestyle With Occupational Therapy for Chronic Pain Patients
Acronym: REVEAL(OT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slagelse Hospital (Other)
Collaborators: University of Southern Denmark (Other); Danish Association of Occupational Therapist (Other); Region Zealand (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Svetlana Solgaard Nielsen, BSc/MSc in Health (Occupational Therapy), Slagelse Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJ-703
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Chronic Pain
Keywords: Activities of daily living; Occupational performance; Quality of life; Health behaviour change; Healthy eating; Physical activity; Occupational Therapy
MeSH Terms: conditions — Chronic Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Adults with chronic pain (n=48) matching the inclusion and exclusion criteria will be included.
  Interventions: Behavioral: Lifestyle-oriented Occupational Therapy added to current treatment of chronic non-malignant pain

INTERVENTIONS:
Behavioral: Lifestyle-oriented Occupational Therapy added to current treatment of chronic non-malignant pain — The participants are recruited from the outpatient cohort admitted at The Multidisciplinary Pain Center (MPC) at Naestved Hospital (Zealand Region, Denmark). The participants receive both, the current treatment based on Cognitive Behavioural Therapy (CBT) and delivered by physicians, nurses, physical therapists and a social worker as usual care, and a lifestyle-oriented Occupational Therapy intervention. The Occupational Therapy intervention targets meaningful daily occupations, physical activity, and eating habits and routines. The intervention is delivered by graduated occupational therapists once á week during the 15 weeks after the initial 5-weeks compulsory psychoeducation course at the MPC. The intervention contains in-person contacts with OTs every other week (e.g. two 1-hour individual sessions at the hospital and/ or at-home and five 2-hours group sessions) and seven phone consultations in the opposite weeks.

SUMMARY:
About 20-30% of the Danish population suffers from chronic non-malignant pain. Current evidence suggests that a bio-psychosocial treatment delivered by multidisciplinary teams is the most effective treatment of chronic non-malignant pain. However, the evidence is still missing on the optimal multimodal treatment combination as well as the additional effect of specific treatment modalities.

A lifestyle-focused intervention is considered to be a relevant supplement to the multidisciplinary treatment of chronic non-malignant pain. Occupational therapy (OT) has previously demonstrated effectiveness in changing the lifestyle of adults through a holistic, systems-based approach. To our knowledge, the method has not previously been approved as a part of the multidisciplinary treatment of adults with chronic non-malignant pain.

The aim of this study is to evaluate the feasibility of the lifestyle-oriented OT intervention added to the current treatment for adults with chronic non-malignant pain, to inform the design and conduct of the future RCT.

DETAILED DESCRIPTION:
Methods

Design

The feasibility study is designed as a mixed-methods single-arm case series pretest-posttest study. The feasibility of the planned intervention course and the assessment procedures will be evaluated. Forty-eight adults aged 18-65 will receive the lifestyle-oriented OT intervention for 15 weeks in addition to the current multidisciplinary CNMP treatment. The participants will complete assessments for Quality of Life (EQ-5D-5L), Occupational performance (COPM, AMPS), Occupational balance (OBQ), Pain-related Self-efficacy (PSEQ), Physical wake-time activity (actigraphs), BMI (weight and height scale), Waist circumference (measuring tape), Blood pressure (sphygmomanometer), and Central pain sensitization at baseline and upon OT intervention discharge. Adverse events (AE) will be registered.

Satisfaction with the add-on OT treatment among the participants and the multidisciplinary team members will be investigated through qualitative research methods. All the steps of the OT intervention will be evaluated by the participants qualitatively and quantitatively throughout the course. Focus group interviews with the participants and the multidisciplinary team inclusive OTs will be conducted upon the end of the OT intervention.

Ethical standards

The feasibility study follows the principles of The World Medical Association (WMA) described in the WMA Declaration of Helsinki. Ethical approval was obtained from the Research Ethics Committeé (SJ-703) and the Data Protection Authority (REG-052-2018) in Zealand Region, Denmark. The feasibility study is conducted in compliance with the European Union's (EU) General Data Protection Regulation (GDPR) and the Danish Data Protection Act.

Recruitment

The participants are enrolled from the outpatient cohort referred to the MPC as usual (e.g. by family physician etc.). All the admitted outpatients are approved for eligibility by a trained project assistant. Detailed written and oral information on the project, and invitation to participate, is provided to the outpatients who meet the inclusion and exclusion criteria. Informed consent on participation is obtained.

Sample

A total of 48 participants is estimated as sufficient for the feasibility study. All the participants are the citizens living in the Zealand Region, Denmark.

Intervention

The participants attend a lifestyle-oriented OT intervention combined with the current treatment at the MPC. The current treatment at the MPC may include medication adjustments, consultation, education, exercises, and homework, with Cognitive Behavioural Therapy (CBT) being the major approach. The patients start the treatment course with a 5-weeks (1,5 hour á week) compulsory group-based psychoeducation course delivered by the MPC's health professionals, e.g. physicians, nurses, physiotherapists, psychologists, and a social worker. The treatment continues afterward as individual treatment sessions by relevant health professionals. Every individual treatment composition is agreed upon by the patient and the multidisciplinary team. Group treatments are available through the MPC's Pain School, mindfulness course, positioning group course, pain treatment group for men and fibromyalgia group for women. The transcutaneous electrical nerve stimulation (TENS) is offered when relevant.

A lifestyle-oriented OT intervention is developed to complement the current treatment at the MPC. Inspired by the Lifestyle Redesign®-concept (USA), the OT intervention includes client-centered education, peer exchange, personal reflection and practicing in-vivo. The OT intervention is delivered by graduated OTs during the 15 weeks and runs parallel with the individual treatment at the MPC, after the psychoeducational course. The OT intervention has a three-fold focus on meaningful daily occupations, physical activity, and eating habits and routines. The OT intervention provides outpatients with an OT contact once a week, in-person every other week and by phone in the opposite weeks. The in-person contacts contain two 1-hour individual sessions and five 2-hours group sessions. One of the in-person individual sessions may be offered as a home visit in terms of an evaluation of home environments, when relevant. The groups are composed of six participants that will meet at the OT Department at Naestved Hospital.

The intervention manual is developed for the study. The trained intervention OTs receive supervision from the project leader during the intervention once a week, or upon demand. Cooperation with the multidisciplinary team at the MPC and inter-sectoral units on local communities across Zealand Region will be provided on an interdisciplinary basis and according to the participant's needs.

Data collection procedures

The project operates with data from patient journals and the Danish quality and research database PainData (approved by The Danish Data Protection Agency as a quality and research database, Reg. nr. 14/44319). The original questionnaire in PainData is supplied with additional questions for the specific project needs. Upon the recruitment and before the baseline assessment, the participants receive electronic access to the PainData and fill in the questionnaire. Thus, demographic and pain-related data, self-reported Quality of Life (QoL), Occupational balance, Pain Self-efficacy, and AE are registered in PainData.

After being admitted to the MPC and recruited to the project, the participants meet for the baseline assessment round that varies 2,5 hours, inclusive breaks. The participants complete the assessment of Occupational performance, Weight, Height, Waist circumference, Blood pressure, and Central sensitization. The participants are provided actigraphy-units (actimetry sensors) for home monitoring of rest-activity cycles. Detailed instructions for home monitoring is provided. The post-discharge assessment round follows the same procedure and is carried out after the ended OT intervention, approximately 5-6 months from the treatment start at the MPC.

The assessment of Occupational performance is performed by graduated OTs with appropriate qualifications. Physical wake-time activity cycles are obtained as self-assessment. Adherence to treatment is assessed by the registration of sessions attended or missed by each participant. Phone calls are used to establish compliance and prevent missing data. Qualitative data from the interviews are collected and transcribed. The transcription process is conducted by two undependable researchers.

Measures

The outcome measures in this trial are based on the recommendations for chronic pain clinical trials from the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) and include the core chronic pain outcome domains, such as participants' rating of overall improvement, pain intensity, physical functioning, and emotional functioning. Validated OT tools investigating occupational performance and balance will be included. The monitoring of lifestyle parameters and activity levels is conducted. Demographic characteristics allow the detection of potential confounders.

Adverse Events

Adverse events (AE) are defined as undesirable experiences during follow-ups, such as death, life-threatening disease, hospitalization, disability or permanent damage (or any need for prevention of those), and other serious health issues with a need for medical or surgical treatment. AEs are registered in the generic questionnaire in the Danish quality and research database PainData. Those untimely discontinued from the study receive a phone call in terms of the discontinuation causes. For all AEs, the date of occurrence, duration, and potential consequences are assessed.

The study course does not have any obvious risks of adverse effects for the participants. Any possible risks for the participants can be considered as minimal and unlikely, while multiple benefits will be expected, for both the actual and the future CNMP-patients. By an injury, the patients are able to seek the Patient Compensation.

Analysis

Data analysis will inform further decisions on a subsequent randomized controlled trial and adjustments in the OT intervention, and improvements of the multidisciplinary team cooperation during a treatment course. Explorative analysis of quantitative and qualitative data will examine the possible effects of the intervention and shortcomings. Whether the study population is normally distributed or not, quantitative methods, such as paired-samples t-test or Wilcoxon signed-rank test, will be used to estimate gain scores from the treatment.

Qualitative data will be analyzed through the following steps to ensure rigorous analysis of the qualitative data: i) mutual coding manual developed during the coding process; ii) iterative coding process where similarities and differences will be identified; iii) research group discussion and agreement during the analysis process; and iv) triangulation of quantitative and qualitative data on acceptability and satisfaction by the treatment.

Dissemination

All the significant, non-significant and/ or inconclusive results will be explicated and published.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18<65yr, chronic non-malignant pain diagnosis present ≥ 3 mths at the inclusion

Exclusion Criteria:

* Acute/ sub-acute pain; cancer-related pain; unstable medicine intake over the past four weeks; daily opioid intake >30 mg; headache/migraine; currently diagnosed depression; current substance misuse; severe psychiatric diagnosis; poor Danish speaking skills and participating in other CNMP-treatment programs. Severe psychiatric diagnoses are defined as a mental illness involving distortion in thinking and perception, and leading to significant social and occupational dysfunction, e.g. schizophrenia and schizotypal, delusional, schizoaffective or psychotic disorders, or psychosis.

Both, new eligible patients, and those who fulfill the eligibility criteria after an initial opioid intake adjustment course, will be considered.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life (EQ-5D-5L Index) from baseline to post discharge | Baseline and 6 months from baseline
  The participants will evaluate their subjective health state in domains Mobility, Self-care, Usual activities, Pain/ Discomfort and Anxiety/ Depression on a 5-point Likert scale from 1= having no problems, having slight problems, having moderate problems, having severe problems and 5= being unable to do/having extreme problems.

SECONDARY OUTCOMES:
Change in Occupational Performance and satisfaction from baseline to post discharge | Baseline and 6 months from baseline
  Obtained by The Canadian Occupational Performance Measure (COPM), Self-reported The COPM is an interview-based OT tool that measures occupational performance in all areas of life and throughout different life stages. The COPM will help the client to identify the issues related to self-care, leisure and productivity, to assess a degree of importance of those for the individual, to prioritize the occupational issues, and to detect changes in self-perceived occupational performance from one point of time to another. The COPM will provide basis for setting intervention goals.
Change in Motor and Process Skills from baseline to post discharge | Baseline and 6 months from baseline
  Obtained by The Assesment of Motor and Process Skills (AMPS), Observed The AMPS is an OT tool that helps to evaluate the overall ability to perform domestic or instrumental activities of daily living (ADL), as well as motor and process skills, in an individual. Motor skills are defined as the observable actions that have been made by an individual during an ADL-performance. Process skills are defined as the observable operations, an individual has made in terms of organizing and proceeding his or her occupational performance.
Change in Occupational balance from baseline to post discharge | Baseline and 6 months from baseline
  The Occupational Balance Questionnaire, Danish version (OBQ-DK), Self-reported The OBQ is an OT-tool that consists of 13 items and six-steps ordinal scales (from 1 to 4; min. 13 - max. 52) expressing certain amount and variation of occupation in an individual, and defining personal satisfaction with those. A higher score means a better outcome.
Change in Pain Self-efficacy from baseline to post discharge | Baseline and 6 months from baseline
  Obtained by Pain Self Efficacy Questionnaire (PSEQ), Self-reported The PSEQ is a 10-item (0-6 scores; min. 0 - max. 60) questionnaire that helps to assess how confident an individual is with his or her activity performance, e.g. household chores, socializing and work, while in pain. The PSEQ can be applied to all pain presentations. A higher score means a better outcome.
Change in Physical wake-time activity from baseline to post discharge | Baseline and 6 months from baseline
  Obtained by actigraphy units (actimetry sensors) all around the day (24 hours) in 4 days To monitor rest-activity cycles, and thus everyday amount of physical activity, actimetry sensors will be worn by the participants for a period of four days
Change in BMI from baseline to post discharge | Baseline and 6 months from baseline
  Weight and height measures will be obtained by not-wearing shoes or heavy clothes Considering the evidence on common presence of co-morbid obesity in chronic pain conditions, the BMI will be measured by validated weight scale (Tanita DC-360S) and height scale (SECA), to monitor weight changes throughout the intervention. The BMI is defined as a person's weight in kilograms divided by the square of the person's height in meters (kg/m2).
Change in Waist circumference from baseline to post discharge | Baseline and 6 months from baseline
  Obtained by a measuring tape (SECA) WC will be measured by measuring tape wrapped around the waist, parallel to the floor and not twistet, with one layer of thin clothes between the body and the measuring tape, and the bottom edge of the measuring tape aligned with the top of the hip bone. WC as the specific measure to detect the amount of abdominal fat, is found to effectively support BMI assessment and identify the risk of metabolic syndrome in a person.
Change in Blood pressure from baseline to post discharge | Baseline and 6 months from baseline
  Obtained by Sphygmomanometer (MicroLife BPA3L Comfort) According to the evidence, chronic pain may cause hypertension, and thus, higher cardio-metabolic risks. BP was measured by a sphygmomanometer, with an inflatable rubber cuff wrapped around the left arm.

OTHER OUTCOMES:
Change in Quantitative sensory testing (QST) for somatosensory pain perception | Baseline and 6 months from baseline
  Controlled Cuff Pressure Algometry (CCPA) unit, with two cuffs applied under the knees CCPA will be used in the study as a standardized QST method is applicable to various chronic pain conditions and able to identify general pain sensibility in an individual, based on deep tissue somatosensory pain response. To minimize the assessment load, other QST methods will not be used in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette R. Christensen, OT, PhD, Principal Investigator — Department of Public Health, University of Southern Denmark; Soeren T. Skou, PT, PhD, Study Director — Slagelse Hosp.; Dept. of Sports Science & Clin. Biomechanics, Univ. of South. DK
Locations (1):
- Naestved, Slagelse and Ringsted Hospitals, Slagelse, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen SS, Skou ST, Larsen AE, Polianskis R, Arendt-Nielsen L, Ostergaard AS, Kjaer-Staal Petersen K, Vaegter HB, Sondergaard J, Christensen JR. Changes in pain, daily occupations, lifestyle, and health following an occupational therapy lifestyle intervention: a secondary analysis from a feasibility study in patients with chronic high-impact pain. Scand J Pain. 2023 Dec 1;24(1). doi: 10.1515/sjpain-2023-0043. eCollection 2024 Jan 1. PMID 38037749
- [Derived] Nielsen SS, Skou ST, Larsen AE, Polianskis R, Pawlak WZ, Vaegter HB, Sondergaard J, Christensen JR. Occupational therapy lifestyle intervention added to multidisciplinary treatment for adults living with chronic pain: a feasibility study. BMJ Open. 2022 Sep 17;12(9):e060920. doi: 10.1136/bmjopen-2022-060920. PMID 36115674